CLINICAL TRIAL: NCT04063696
Title: AntibaCterial presCribing & OraL Health Practice: The Leeds Dental Extraction Study
Brief Title: AntibaCterial presCribing & OraL Health Practice
Acronym: ACCOLaDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: Oral and Dental Research Trust (Unknown)
Responsible Party: Principal Investigator, Sue Pavitt, Professor in Applied Health and Translational Research, University of Leeds
Other Study IDs: DT17/103574; 231858 (Other: IRAS); 18-WS-0111 (Other: Research Ethics Committee)
Record Dates: First submitted 2018-11-08; First posted 2019-08-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Dental Anxiety; Tooth Loss
Keywords: tooth extraction; dental anxiety; antibiotic; oral health
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study by Allied Health Professionals to explore the experience of patients undergoing tooth extraction at Leeds Dental Institute in relation to antibiotic medication, dental anxiety and oral health practices

DETAILED DESCRIPTION:
Consented patients attending the Leeds Dental Institute for tooth extraction will be asked to complete 3 questionnaires in order for the researchers to understand more about the background of patients who have teeth extracted at the centre. The study will focus on the patient's previous experience of dentistry such as whether they have had antibiotics prescribed for toothache, whether they suffer from dental anxiety and how they regularly look after their oral health.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing extraction of one or more teet
* Parents/Guardians of children aged 5-12 years old undergoing extraction of one or more teeth
* Patients aged 13-15 undergoing extraction of one or more teeth
* Patients and Parents/Guardians who are willing to give informed consent or assent to complete questionnaires

Exclusion Criteria:

* Patients, parents/guardians unable or unwilling to provide informed consent
* Parents/Guardians of patients aged less than 5 years old
* Patients or parents who are unable to communicate directly with the health person carrying out the treatment

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending Leeds Dental Institute for tooth extraction.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-08-23 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Main endpoint: WHO Oral Health Questionnaire for Adults (Annexe 7) or WHO Oral Health Questionnaire for Children (Annexe 8) | Up to 2 hours before tooth extraction procedure
  The use of these two simplified structured questionnaires is recommended by WHO for the collection of self-assessed data on oral health and risk factors in adults (Annex 7) and in children or adolescents (Annex 8). The simplified questionnaires include the core questions considered essential in national oral health surveillance. Complete analysis of answers to the questions on oral health related quality of life, consumption of sugary foods and drinks, consumption of tobacco, and harmful use of alcohol will require derivate variables. There are corresponding questions in the questionnaire to children. Behavioural indices may be generated from these questions by addition of the item scores chosen by the respondent. Cut-off points for categories (3 or 5) may then be determined from empirical distributions.
Main endpoint: Antimicrobial survey | Up to 2 hours before tooth extraction procedure
  Antimicrobial survey
Main endpoint: Modified Child Dental Anxiety Scale (MCDAS) v1.0 dated 17/10/2016 (Wong et al 1998) | Up to 2 hours before tooth extraction procedure
  Modified Child Dental Anxiety Scale (MCDAS) v1.0 dated 17/10/2016 (Wong et al 1998). An 8-question Modified Child Dental Anxiety Scale to assess children's concerns about specific dental procedures, such as dental examination, scale and polish, injection, filling, extraction, and relative and general anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Pavitt, PhD, Study Director — University of Leeds
Locations (1):
- Leeds Dental Institute, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT04063696/Prot_000.pdf